CLINICAL TRIAL: NCT06513078
Title: The Effect of Different Types of Cupping Therapy on Acute Changes in Ankle Dorsiflexion
Brief Title: Different Types of Cupping Therapy and Ankle Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-22-1287
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Ankle dorsiflexion; Dynamic cupping; Static cupping

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants did not know whether they were receiving actual cupping treatment or a sham treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Static cupping (Experimental): Negative pressure was created inside 4 plastic cups (2" diameter) placed on the gastrocnemius by drawing out air with two full pumps via a manual suction tool and participants laid in the prone position for 10 minutes while the cups stayed attached to the skin. Cups were attached to the skin with adhesive tape.
  Interventions: Other: Static cupping
- Static sham cupping (Sham Comparator): Negative pressure was created inside 4 plastic cups (2" diameter) placed on the gastrocnemius by drawing out air with two full pumps via a manual suction tool and participants laid in the prone position for 10 minutes while the cups stayed attached to the skin. Cups were attached to the skin with adhesive tape. However, the sham cups had a small hole in them which allowed pressure to leak out.
  Interventions: Other: Static sham cupping
- Dynamic cupping (Experimental): Negative pressure was created inside 4 plastic cups (2" diameter) placed on the gastrocnemius by drawing out air with two full pumps via a manual suction tool and participants laid in the prone position for 5 minutes while the cups stayed attached to the skin. Participants then completed two sets of 10 full range ankle pumps with a rest period of 30 seconds between sets (approximately 2 minutes). For the remaining 3 minutes, participants remained still in the prone position with the cups remaining attached. Cups were attached to the skin with adhesive tape.
  Interventions: Other: Dynamic cupping
- Dynamic sham cupping (Sham Comparator): Negative pressure was created inside 4 plastic cups (2" diameter) placed on the gastrocnemius by drawing out air with two full pumps via a manual suction tool and participants laid in the prone position for 5 minutes while the cups stayed attached to the skin. Participants then completed two sets of 10 full range ankle pumps with a rest period of 30 seconds between sets (approximately 2 minutes). For the remaining 3 minutes, participants remained still in the prone position with the cups remaining attached. Cups were attached to the skin with adhesive tape. However, the sham cups had a small hole in them which allowed pressure to leak out.
  Interventions: Other: Dynamic sham cupping

INTERVENTIONS:
Other: Static cupping — 4 cups were placed on the gastrocnemius, negative pressure was applied and participants lay prone on a table for 10 minutes.
  Arms: Static cupping
Other: Static sham cupping — 4 cups were placed on the gastrocnemius, negative pressure was applied and participants lay prone on a table for 10 minutes. A pin hole in the cup allowed pressure to slowly leak out during the treatment.
  Arms: Static sham cupping
Other: Dynamic cupping — 4 cups were placed on the gastrocnemius, negative pressure was applied and participants lay prone on a table for 5 minutes, then did ankle exercises for 3 minutes, and lastly lay prone on the table for the last 3 minutes.
  Arms: Dynamic cupping
Other: Dynamic sham cupping — 4 cups were placed on the gastrocnemius, negative pressure was applied and participants lay prone on a table for 5 minutes, then did ankle exercises for 3 minutes, and lastly lay prone on the table for the last 3 minutes. A pin hole in the cup allowed pressure to slowly leak out during the treatment.
  Arms: Dynamic sham cupping

SUMMARY:
The purpose of this study was to determine the acute effects of different manual cupping therapy protocols on ankle range of motion, compared to sham treatments, in generally healthy adults with limited ankle range of motion (i.e., ankle dorsiflexion less than 40 degrees).

DETAILED DESCRIPTION:
The purpose of this study was to determine the acute effects of different manual cupping therapy protocols on ankle range of motion, compared to sham treatments, in generally healthy adults with limited ankle range of motion (i.e., ankle dorsiflexion less than 40 degrees). Participants had their baseline ankle dorsiflexion measured with a digital inclinometer in a weight-bearing modified lunge position by a certified athletic trainer. Participants who were eligible for the study were then randomly assigned to one of 4 groups; 2 of which were intervention groups (i.e., dynamic cupping, static cupping) and 2 of which were sham treatments (i.e., static sham cupping, dynamic sham cupping). Each participant was blinded to the therapy they were randomized to and all received a total of 10 minutes of the cupping therapy (either actual or sham). In general, cupping therapy consisted of creating a negative pressure in four 2" diameter plastic cups placed on the gastrocnemius. Sham cups had small holes in them allowing air to leak out. Cups were also attached with adhesive tape to all participants to ensure blinding. Depending on the treatment received, participants either were asked to lie still in the prone position or perform ankle exercises during the 10 minutes while the cups were attached. Immediately after receiving treatment, participants had their ankle dorsiflexion measured again using the same procedure described for baseline measurement.

ELIGIBILITY:
Inclusion Criteria:

* Limited ankle dorsiflexion (less than 40 degrees of weight bearing ankle dorsiflexion at baselines)
* Never received cupping therapy prior to the study
* No lower extremity injuries in the past 6 months
* No contraindications associated with cupping therapy (e.g., deep vein thrombosis, pregnancy, bone fracture, or sunburn/rash)
* Generally healthy

Exclusion Criteria:

* Ankle dorsiflexion greater than or equal to 40 degrees during weight bearing ankle dorsiflexion at baseline
* Received cupping therapy in the past
* Has a lower extremity injury or has had a lower extremity injury in the past 6 months
* Self-reported a contraindication associated with cupping therapy (e.g., deep vein thrombosis, pregnancy, bone fracture, or sunburn/rash).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in average ankle dorsiflexion (degrees) using a digital inclinometer | Baseline and immediately after receiving treatment.
  Weight bearing ankle dorsiflexion measured by performing a modified lunge and bringing the knee forward as far as possible without allowing the heel to come off of the ground. A digital inclinometer was placed vertically over the tibial tuberosity and the measurement was reported as the average of three trials, in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Megan C Nelson, PhD, Principal Investigator — Northern Michigan University
Locations (1):
- Northern Michigan University, Marquette, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared, data will only be shared in aggregate form.